CLINICAL TRIAL: NCT04382885
Title: Pharmacokinetics, Safety, and Tolerability of Cariprazine in Pediatric Participants With Autism Spectrum Disorder Aged 5-17 Years
Brief Title: Cariprazine Pediatric ASD PK Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000-103-009
Record Dates: First submitted 2020-03-19; First posted 2020-05-11 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — cariprazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (10-17 years) (Experimental): 10 to 12 years: 0.75 mg/day cariprazine oral solution 13 to 17 years: 1.5 mg/day cariprazine oral solution
  Interventions: Drug: Cariprazine
- Cohort 2 (10-17 years) (Experimental): 10 to 12 years: 1.5 mg/day cariprazine oral solution 13 to 17 years: 3.0 mg/day cariprazine oral solution
  Interventions: Drug: Cariprazine
- Cohort 3 (5-9 years) (Experimental): 0.5 mg/day cariprazine oral solution
  Interventions: Drug: Cariprazine
- Cohort 4 (5-9 years) (Experimental): 1.5 mg/day cariprazine oral solution
  Interventions: Drug: Cariprazine

INTERVENTIONS:
Drug: Cariprazine — Oral Solution

SUMMARY:
This study will be a multi-center, open-label, parallel-group, multiple-dose study in up to 24 male and female participants aged 5 through 17 years, inclusive, with Autism Spectrum Disorder (ASD). The 24 participants will be enrolled into 1 of 4 cohorts (6 participants per cohort).

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) criteria for ASD (Autism Spectrum Disorder) diagnosis.
* Participants must have normal physical examination findings and clinical laboratory test results for their age group or abnormal results judged not clinically significant by the investigator.
* Negative serum hCG (human chorionic gonadotropin) pregnancy test at screening (all female participants that have reached menarche).
* BMI greater than the 5th percentile for age and gender based on CDC (Centers for Disease Control and Prevention) growth charts.
* Participant (if reached his spermarche or her menarche), must agree to sexual abstinence or to use an approved birth control method for the full duration of participation in the study. The investigator and each participant will determine the appropriate method of contraception for the participant during their participation in the study.
* Participant's parent(s)/legal representative(s) must be capable of giving signed informed consent , which includes compliance with the requirements and restrictions listed in the ICF and in the protocol as explained by the investigator. Written informed consent from the participant's parent(s)/legal representative(s) must be obtained prior to any study-related procedures.
* Assent (unless local regulations require consent) must be obtained for all participants participating in the study.
* Participant must have a parent or legal representative who is willing and able to be responsible for safety monitoring of the participant, provide information about the participant's condition, oversee administration of study intervention, and accompany the participant to all study visits. The caregiver can be the participant's parent(s)/legal representative(s). Written consent from the caregiver must be obtained.

Exclusion Criteria:

* Current diagnosis of bipolar disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, brief psychotic disorder, or psychotic disorder due to another medical condition.
* Diagnosis of intellectual disability (IQ < 70) documented by school record, neuropsychological testing or medical records.
* Participant has a history of meeting DSM-5 diagnosis for any substance-related disorder (except caffeine- and tobacco-related) within the 3 months before the Screening Visit.
* Participant with an acute or unstable medical condition, including (but not limited to) inadequately controlled diabetes, hepatic insufficiency (specifically any degree of jaundice), uncorrected hyper- or hypo-thyroidism, acute systemic infection, renal, gastrointestinal, respiratory, or cardiovascular disease.
* History of seizures, with the exception of febrile seizures.
* History of tumor of the central nervous system.
* Previously taken cariprazine or previously participated in an investigational study of cariprazine.
* Participant is currently enrolled in an investigational drug or device study or participation in such a study within 3 months of Study Day 1.
* Participation in a blood or plasma donation program within 60 or 30 days, respectively, prior to Study Day 1.
* Positive UDS for substances of abuse at the Screening Visit or on Study Day -1.
* Known allergy or sensitivity to the study intervention or its components.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 30 days after last visit or last dose for participants who discontinue early
Incidence of Serious Adverse Events (SAEs) | Up to 30 days after last visit or last dose for participants who discontinue early
Incidence of AEs leading to discontinuation | Up to 30 days after last visit or last dose for participants who discontinue early
Percentage of participants with potentially clinically significant values in clinical laboratory assessments | Up to 84 days
Percentage of participants with potentially clinically significant values in vital signs assessments | Up to 84 days
Percentage of participants with potentially clinically significant values in ECG assessments | Up to 84 Days
Percentage of participants who have suicidal ideation or suicidal behaviors in C-SSRS assessments | Up to 84 Days
Percentage of participants with treatment-emergent parkinsonism in SAS assessments | Up to 84 Days
Percentage of participants with treatment-emergent akathisia in BARS assessments | Up to 84 days
Percentage of participants with potentially clinically significant values in ocular examination parameters | Screening to Day 84
Pharmacokinetics: Maximum plasma concentrations (Cmax) of cariprazine and its metabolites DCAR and DDCAR on Days 1 and 42 | Day 1 and Day 42
Pharmacokinetics: Time of maximum plasma concentrations (Tmax) of cariprazine and its metabolites DCAR and DDCAR on Days 1 and 42 | Day 1 and Day 42
Pharmacokinetics: Area under the plasma concentration-time curve during the dosing interval (AUC0-tau) of cariprazine and its metabolites DCAR and DDCAR on Days 1 and 42 | Day 1 and Day 42
Pharmacokinetics: Terminal elimination half-life (T1/2) of cariprazine and its metabolites DCAR and DDCAR | Day 42 to Day 84
Pharmacokinetics: Minimum plasma concentrations (Cmin) during the dosing interval of cariprazine and its metabolites DCAR and DDCAR on Day 42 | Day 42
Pharmacokinetics: Average plasma concentrations (Cavg) during the dosing interval of cariprazine and its metabolites DCAR and DDCAR on Day 42 | Day 42
Pharmacokinetics: Apparent total clearance of cariprazine from plasma (CL/F) on Day 42 | Day 42
Pharmacokinetics: Volume of distribution during the terminal elimination phase (Vz/F) of cariprazine | Day 42 to Day 84

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (3):
- United States (3):
  - Neuropsychiatric Research Center of Orange County /ID# 233663, Orange, California
  - Atlanta Center for Medical Research /ID# 233576, Atlanta, Georgia
  - iResearch Atlanta, LLC /ID# 233614, Decatur, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. — http://www.AllerganClinicalTrials.com
- See also: To be considered as a site for current and future Allergan Clinical Trials, please register using the Investigator Databank link. — http://www.investigatordatabank.org/